CLINICAL TRIAL: NCT00024375
Title: Phase II Open-Label Study of Taxoperxin (DHA-Paclitaxel) Injection by 2 Hour Intravenous Infusion in Patients With Metastatic Cancer of the Pancreas
Brief Title: DHA-Paclitaxel in Treating Patients With Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068926; THERADEX-P01-00-03; PROTARGA-P01-00-03; VMRC-8770
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2003-03

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — docosahexaenoyl-paclitaxel

INTERVENTIONS:
Drug: DHA-paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DHA-paclitaxel in treating patients who have metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tumor response rate, duration of response, and time to disease progression in patients with metastatic carcinoma of the pancreas treated with DHA-paclitaxel.
* Determine the overall survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.
* Assess the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive DHA-paclitaxel IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 2 courses, and at completion of treatment.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma of the pancreas

  * Metastatic disease
* Measurable disease

  * Lesions within a previously irradiated field are not considered measurable
* No islet cell tumors, lymphoma, or sarcoma of the pancreas
* No known or clinical evidence of CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled ventricular arrhythmia
* No myocardial infarction within the past 3 months
* No superior vena cava syndrome

Neurologic:

* No peripheral neuropathy greater than grade 1
* No uncontrolled major seizure disorder
* No spinal cord compression

Other:

* No concurrent serious infection requiring parenteral therapy
* No unstable or serious concurrent medical condition
* No other prior malignancy except:

  * Curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix OR
  * Other cancer curatively treated with surgery alone that has not recurred for more than 5 years
* No psychiatric disorder that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy for metastatic disease
* Prior adjuvant chemoradiotherapy allowed
* At least 28 days since prior chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except megestrol

Radiotherapy:

* See Disease Characteristics
* Prior adjuvant chemoradiotherapy allowed
* At least 28 days since prior large-field radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 14 days since prior major surgery and recovered

Other:

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (4):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- Germany (2):
  - Kliniken Essen - Mitte, Essen
  - Krankenhaus Nordwest, Frankfurt
- Erasmus Medical Center, Rotterdam, Netherlands
- United Kingdom (2):
  - New Cross Hospital, Wolverhampton, England
  - Beatson Oncology Centre, Glasgow, Scotland